CLINICAL TRIAL: NCT03573713
Title: Decreasing Stunting by Reducing Maternal Depression in Uganda - A Cluster Randomized Controlled Trial (CRCT) for Improved Nutrition Outcomes
Brief Title: Decreasing Stunting by Reducing Maternal Depression in Uganda: A Cluster Randomized Controlled Trial (CRCT) for Improved Nutrition Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food for the Hungry (Other)
Collaborators: Teachers College, Columbia University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Godfrey Opiyo, FH Uganda ECF Program Coordinator, Food for the Hungry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FHU-ECF
Record Dates: First submitted 2018-03-15; First posted 2018-06-29 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Depression, Postpartum; Malnutrition, Child
Keywords: Hygiene practices; Sanitation; Nutrition; Interpersonal Psychotherapy; Maternal depression; clustered randomized controlled trial
MeSH Terms: conditions — Depression, Postpartum; Child Nutrition Disorders | interventions — Interpersonal Psychotherapy; Population Groups

STUDY DESIGN:
Intervention Model Description: IPT-G Promoters will screen all women for depression who are pregnant or will have a child who will be 18m old or younger by 2 May 2018 in each of the 34 Care Group Service Areas chosen for the study. If informed consent is obtained and the women's scores on the PHQ-9 indicate mild to severe depression, they will be put into groups of approx. 8 women for IPT-G. The 34 Care Group Service Areas (CGSAs) will then be randomized into 2 arms (IPT-G and control). Women in the CGSAs in the IPT-G arm who screen positive for depression will receive IPT-G for 12 weeks. Following IPT-G treatment, all women who are pregnant or that have a child born on or after 3 August 2016 in the project area will be provided with psychoeducation through the Care Group structure. For the assessments conducted after the baseline, trained external (non-staff) enumerators will be used to assess for depression and other things, and they will be blind to which group the mothers are in (treatment or control).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPT-G (Treatment arm) (Experimental): This arm will receive IPT-G for 12 weeks. Following IPT-G, this arm will go on to receive the Care Group intervention parallel to the control arm.
  Interventions: Behavioral: IPT-G
- Control arm (Treatment as usual - Care Group) (Other): This arm will receive assessment only at the beginning of the study (parallel to the start of IPT-G) and then receive the Care Group intervention after 12 weeks together with the IPT-G arm.
  Interventions: Other: Care Groups

INTERVENTIONS:
Other: Care Groups — The Care Groups model has strong evidence of improvement of maternal and child health and maternal hygiene/nutrition behaviors.Through Care Groups, women will learn about proper water, sanitation, and hygiene behaviors; Infant and Young Child Feeding practices; management of childhood illnesses; home management, referral and care seeking for sick children; family planning; and use of preventive services available at health facilities (e.g., growth monitoring, deworming, vitamin A supplementation). All children under five years of age will also be screened for acute malnutrition by the Care Group Volunteers, and receive deworming medication and vitamin A supplementation twice a year through the Ministry of Health and Community Health Workers as part of national campaigns.
  Other Names: CG
  Arms: Control arm (Treatment as usual - Care Group)
Behavioral: IPT-G — IPT-G is an effective, low-cost, short-duration community-based method for decreasing depression has been established that was first rigorously tested in Uganda. Several Private Voluntary Organizations in Africa have used this low-cost, short-duration, community-based group psychosocial approach and found it to be a culturally-sensitive, acceptable, and feasible approach to address depression.
  IPT-G treatment spans 12 weeks of treatment, consisting of 3 phases (early, middle, and termination). Within this treatment, participants are also assessed for symptoms of depression every week.
  Other Names: Interpersonal Psychotherapy for Groups
  Arms: IPT-G (Treatment arm)

SUMMARY:
The project seeks to test the integration of Interpersonal Psychotherapy for Groups within Care Group projects and investigate whether the treatment of maternal depression with Interpersonal Psychotherapy for Groups improves the adoption of nutrition-related behaviors that can reduce stunting in the Kitgum District in northern Uganda. A secondary aim is to examine whether the participation in the care groups will also result in remission of depression as a non-specific therapeutic effect although it may not be intended as an antidepressant treatment.

DETAILED DESCRIPTION:
Over the past two decades there has been a growing global momentum and commitment to address malnutrition. The most recent indication of this is reflected in goal #2 of the Sustainable Development Goals, "end hunger, achieve food security and improved nutrition and promote sustainable agriculture." However, great challenges remain. Today, over 165 million children under five are chronically malnourished or stunted, and once a child is stunted, it is nearly impossible to regain their cognitive and physical potential. In addition, it is estimated that malnutrition contributes to more than one-third of all child deaths under the age of five.

Through research and fieldwork, key evidence-based interventions and target populations have been identified. It has been found that the most critical time to prevent chronic malnutrition is from conception up through the child's second birthday, known as the "first 1,000 days." Improving household behaviors related to maternal and child health and nutrition such as improved water, sanitation, and hygiene practices, proper infant and young child feeding practices, optimal maternal nutrition and antenatal care, and others can reduce child malnutrition and prevent up to 57% of deaths of children under five years of age.

However, despite the gains in reducing stunting in children, there has been no program implemented at scale that has come close to normalizing child growth. There is a need for new tools and interventions that focus on other causes of malnutrition aside from poor water, sanitation, and hygiene, infant and young child feeding, home management/care seeking for sick children, maternal nutrition/antenatal care, and use of preventive services (e.g., immunizations). One promising new intervention is the treatment of maternal depression, an underlying cause of malnutrition. The potential global impact of adding community-based treatment of maternal depression to the investigator's toolbox of interventions to reduce child stunting could be significant: A recent meta-analysis found that stunting could be reduced globally by about 27% by eliminating maternal depression (Surkan, J, Kennedy C, Hurley, B, and Black, M., 2011). As such, the investigators believe that treatment of maternal depression could result in improved nutrition behavior change in mothers, leading to significant reductions in child stunting and helping to end hunger.

An effective, low-cost, short-duration community-based method for decreasing depression has been established that was first rigorously tested in Uganda: Interpersonal Psychotherapy for Groups. Several Private Voluntary Organizations in Africa have used this low-cost, short-duration, community-based group psychosocial approach and found it to be a culturally-sensitive, acceptable, and feasible approach to address depression. A cluster randomized controlled trial of this approach in depressed adults in southern Ugandan rural communities yielded a 93% decline in diagnosable depression (vs. a 45% decline in controls), as well as significantly higher functionality in household tasks, including those associated with child nutrition and health (Bass et al, 2006). However, this study did not measure changes in maternal adoption of behaviors that affect child nutritional status and the possible effect of treatment of maternal depression on improved child growth. Demonstrating that Interpersonal Psychotherapy for Groups works for increasing maternal adoption of behaviors that affect child nutritional status could have a profound effect on how malnutrition is prevented worldwide, and save children and their mothers from a lot of unnecessary suffering.

Therefore, Food for the Hungry in partnership with the team at the Global Mental Health Lab at Teachers College, Columbia University is proposing a 33 month project which will test how to integrate Interpersonal Psychotherapy for Groups within Care Group projects and whether the treatment of maternal depression with Interpersonal Psychotherapy for Groups improves the adoption of maternal behaviors that can reduce stunting in Kitgum District in northern Uganda. Using a cluster randomized controlled trial design, Food for the Hungry will test whether adding Interpersonal Psychotherapy for Groups for half of the women identified with depression improves the adoption of household health and nutrition behaviors known to improve child linear growth.

Pregnant women and mothers with a child born after 3 April 2016 (who will be under 18 months of age by the time health promotion begins on 4 October 2017) will be assessed for depression, and half of those who meet a cutoff for depression will be randomly assigned to IPT-G. Following the three-month implementation of Interpersonal Psychotherapy for Groups, all pregnant women and women with children under two years of age in the project area will participate in Care Groups, an evidence-based community nutrition promotion model to improve maternal and child health and nutrition behaviors. A recent set of papers summarized the history of Care Groups and the outcomes achieved with the model on children under two years of age in many countries around the world (Perry et al, 2015), and how projects using Care Groups are achieving on average more than double the behavior change of other models on maternal behaviors that affect the growth of children 0-23m (George et al, 2015). Through Care Groups, women will learn about proper water, sanitation, and hygiene behaviors; Infant and Young Child Feeding practices; management of childhood illnesses; home management, referral and care seeking for sick children; family planning; and use of preventive services available at health facilities (e.g., growth monitoring, deworming, vitamin A supplementation). All children under five years of age will also be screened for acute malnutrition by the Care Group Volunteers, and receive deworming medication and vitamin A supplementation twice a year through the Ministry of Health and Community Health Workers as part of national campaigns. Care group experts report improvement of depression as a result of these focus groups, due to the connection, social support and problem-solving among the group members. At the conclusion of this project, a Lessons Learned conference will be held in Uganda and an online dissemination event will be held in order to facilitate the sharing of project results. Results will also be disseminated through peer-reviewed papers and communities of practice.

ELIGIBILITY:
Inclusion Criteria:

* Our study will only include depressed pregnant women and depressed mothers (ages 18 and up) with at least one child under 18 months of age (0-17.9 months) who consent and reside in selected communities in subcounties of Kitgum District of Uganda, as we are aiming to study the effects of the treatment of maternal depression on child care practices during the first few years of life. We will not exclude any classes of subject based on class, race, or ethnicity.

Exclusion Criteria:

* If a woman confirms current risk of suicide or another acute mental health condition (such as psychosis, mania, etc.), she will not be enrolled, but referred to the nearby Peter C. Alderman Kitgum Clinic (Director, Raymond Odonkonyero).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1248 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Change in scores of KPC Survey of maternal and child health and nutrition behaviors | From date of randomization up to 112 weeks. The KPC survey will be administered at three time points: at baseline immediately after randomization; at midpoint (14 weeks after treatment begins), and at termination (at around week 112).
  The "Knowledge, Practices and Coverage" (KPC) survey will measure mothers' endorsement of infant and young child feeding (IYCF) practices; proper water, sanitation, and hygiene (WASH) behaviors; management of childhood illnesses; home management, referral and care seeking for sick children; family planning; and use of preventive services available at health facilities (e.g., growth monitoring, deworming, vitamin A supplementation).

SECONDARY OUTCOMES:
Score of survey on home management, referral and care seeking for children | Around week 26 (end of first CG module)
  * Whether or not mothers of children 0-23m of age who had rapid/difficult breathing or fever in the past two weeks sought care from an appropriate health care provider within 24 hrs of symptoms.
  * Whether or not mothers of children with an illness in the past two weeks gave their child the same/more food or increased breastfeeding in children 0-5m.
  * Whether or not mothers had their child sleep under a long-lasting insecticide-treated net during the past night.
  * Number of signs of childhood illness that require immediately seeking assessment and treatment by a health facility or provider outside of the home known by the mother. (Note: Since these signs of severe illness will affect few children, we are measuring a knowledge indicator here as a proxy for behavior change.)
Score of survey on infant and young child feeding practices | Around week 38 (end of second CG module)
  * Whether or not mothers of children 0-5m are exclusively breastfed and mothers of children 6-23 months of age are giving the child a minimum acceptable diet (apart from breast milk).
  * Whether or not mothers of children 6-23 months of age are giving their child an iron-rich food or iron-fortified food that is specially designed for infants and young children, or that is fortified in the home.
Score of survey on water usage, sanitation and hygiene practices | Around week 47(end of third CG module)
  * Whether or not mothers with children age 0-23 months have soap and water at a hand washing location readily available.
  * Whether or not mothers report proper disposal of the child's feces the last time the child defecated.
  * Whether or not mothers treat household drinking water effectively.
  * Whether or not the mother is depressed.
Score of survey on knowledge and utility of preventive services available at local health facilities | Around week 56 (end of fourth CG module)
  * Whether or not mothers had their child's growth monitored in the past 3 months.
  * Whether or not children 6-24m of mothers received one dose of vitamin A in the past 6m.
  * Whether or not children 9-24m of mothers have received rotavirus vaccine.
Score of survey on family planning practices | Around week 65 (end of fifth CG module)
  ● Whether or not mothers are using an effective method of family planning.

OTHER OUTCOMES:
PHQ-9 | From date of randomization up to 112 weeks. The KPC survey will be administered at three time points: at baseline immediately after randomization; at midpoint (14 weeks after treatment begins), and at termination (at around week 112).
  The 9-Item Patient Health Questionnaire (PHQ-9) assesses an individual for their depression-related feelings and thoughts. The PHQ-9 questions are based on diagnostic criteria of depression from DSM-IV and ask about the patient's experience in the last 2 weeks. Questions are about the level of interest in doing things, feeling down or depressed, difficulty with sleeping, energy levels, eating habits, self-perception, ability to concentrate, speed of functioning and thoughts of suicide. Responses range from "0" (Not at all) to "3" (nearly every day). Clinicians may ask a 10th question that asks how difficult the problems that the prior questions ask about make it to function in daily life. The 10th question is not factored into the final score and clinicians may use it to gauge the patient's opinion of the level of impairment caused by their mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Opiyo, B.S., Principal Investigator — Food for the Hungry; Trisha Okenge, Study Director — Food for the Hungry
Locations (1):
- FH Uganda - Kitgum, Kitgum, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing is pending on sponsor and IRB/data monitoring board approval.

REFERENCES:
- [Background] Surkan PJ, Kennedy CE, Hurley KM, Black MM. Maternal depression and early childhood growth in developing countries: systematic review and meta-analysis. Bull World Health Organ. 2011 Aug 1;89(8):608-15. doi: 10.2471/BLT.11.088187. Epub 2011 May 26. PMID 21836759
- [Background] Bass J, Neugebauer R, Clougherty KF, Verdeli H, Wickramaratne P, Ndogoni L, Speelman L, Weissman M, Bolton P. Group interpersonal psychotherapy for depression in rural Uganda: 6-month outcomes: randomised controlled trial. Br J Psychiatry. 2006 Jun;188:567-73. doi: 10.1192/bjp.188.6.567. PMID 16738348
- [Background] Perry H, Morrow M, Borger S, Weiss J, DeCoster M, Davis T, Ernst P. Care Groups I: An Innovative Community-Based Strategy for Improving Maternal, Neonatal, and Child Health in Resource-Constrained Settings. Glob Health Sci Pract. 2015 Sep 15;3(3):358-69. doi: 10.9745/GHSP-D-15-00051. Print 2015 Sep. PMID 26374798
- [Background] Perry H, Morrow M, Davis T, Borger S, Weiss J, DeCoster M, Ricca J, Ernst P. Care Groups II: A Summary of the Child Survival Outcomes Achieved Using Volunteer Community Health Workers in Resource-Constrained Settings. Glob Health Sci Pract. 2015 Sep 15;3(3):370-81. doi: 10.9745/GHSP-D-15-00052. Print 2015 Sep. PMID 26374799
- [Background] George CM, Vignola E, Ricca J, Davis T, Perin J, Tam Y, Perry H. Evaluation of the effectiveness of care groups in expanding population coverage of Key child survival interventions and reducing under-5 mortality: a comparative analysis using the lives saved tool (LiST). BMC Public Health. 2015 Sep 2;15:835. doi: 10.1186/s12889-015-2187-2. PMID 26329824
- See also: United Nations Sustainable Development Goals — http://www.un.org/sustainabledevelopment/sustainable-development-goals/